CLINICAL TRIAL: NCT04354766
Title: Generation of Human Monoclonal Antibodies Neutralizing SARS-Cov-2 From B Cells of Convalescent Patients
Brief Title: COVID-19 : Neutralizing Human Monoclonal Antibodies Against SARS-Cov-2
Acronym: ANTI-COV-2
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: Eurobio Scientific (Unknown)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_0340; 2020-A01038-31 (Other: ID-RCB)
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: COVID
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Convalescent patients diagnosed with COVID +: Five convalescent patients (minimum 12 days after the onset of symptoms), diagnosed COVID + on the temporary sampling platform that was set up at HCL at the start of the epidemic, which notably concerns symptomatic healthcare professionals for whom hospitalization does not was not necessary.
  Interventions: Other: Blood sample
- Hospitalized convalescent patients diagnosed with COVID +: Five convalescent patients (minimum 12 days after the onset of symptoms), diagnosed COVID +, hospitalized in the infectious diseases department of the Croix-Rousse hospital living in the metropolitan area of Lyon, having presented hypoxaemic pneumonia requiring hospitalization.
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — This study will require a blood sample (4 ACD tubes, 20 ml) at one time.

SUMMARY:
Rationale : The emergence of the novel, pathogenic SARS-coronavirus 2 (SARS-CoV-2) threatens public health. To date, there are no effective drug option to prevent the infection, nor therapeutics for controlling the deadly COVID-19. However, the majority of patients infected with SARS-Cov-2 eliminate the virus by mounting a protective antiviral immune response, associated in particular with the production of neutralizing antibodies. Neutralizing antibodies could be of particular interest for therapeutic purposes, but also for preventive applications, to protect people who have never been in contact with the virus, or immunocompromised patients.

The objectives of this study are :

* To generate human monoclonal antibodies neutralizing SARS-Cov-2 from immortalized B cells of convalescent patients.
* To compare the serological profiles between convalescent patients that develop mild or uncomplicated illness and convalescent patients that develop a more severe disease, that required hospitalization and oxygen support.
* To compare for each patient the neutralizing efficiency of plasma to the neutralizing capacities of the monoclonal antibodies generated with immortalized B cells.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* Patient who signed the study consent form
* Convalescent patient (at least 12 days after the onset of symptoms), having been sampled at Hospices Civils de Lyon for a suspected infection with SARS-Cov-2, confirmed by PCR.

Exclusion Criteria:

* Patient treated with rituximab
* Patient treated with immunoglobulins
* Patient over 18 years old, subject to a legal protection measure (guardianship or trusteeship)
* Patient deprived of liberty
* Pregnant or lactating woman
* Patient not affiliated to a social security scheme or beneficiary of a similar scheme.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study relates to 10 adult subjects who were infected with SARS-Cov-2 (positivity confirmed by PCR test), who were symptomatic, and who were in the recovery phase when the blood sample was collected.
  Among the 10 convalescent subjects who will be sampled, we will select two distinct populations:
  (i) five convalescent patients (minimum 12 days after the onset of symptoms), diagnosed COVID + on the temporary sampling platform which was set up at HCL at the start of the epidemic, which notably concerns symptomatic healthcare professionals for whom hospitalization was not required; (ii) five convalescent patients (minimum 12 days after the onset of symptoms), hospitalized in the infectious diseases department of the Croix-Rousse hospital living in the metropolitan area of Lyon, having presented hypoxemic pneumonia requiring hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2020-04-29 (Actual); Primary Completion 2020-05-18 (Actual); Study Completion 2020-05-18 (Actual)

PRIMARY OUTCOMES:
Production of several human monoclonal antibodies capable of neutralizing the infection of a target cell by SARS-COV-2. | 3 weeks
  Isolation of immortalized B lymphocyte clones, producer of monoclonal antibodies capable of neutralizing the infection of a target cell by SARS-COV-2.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric COUTANT, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital de la Croix-Rousse, Lyon, France